CLINICAL TRIAL: NCT05061186
Title: Effects of Resistive Expiratory Muscle Training on Pulmonary Functions in Patients With COPD Patients
Brief Title: Resistive Expiratory Muscle Training in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01082 Varda Farooq
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: COPD
Keywords: Resistive Expiratory Muscle training; Breathing Exercise; Pulmonary Function; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistive Expiratory muscle Training Group (Experimental): Mild Resistive Expiratory muscle Training Group
  Interventions: Other: Resistive Expiratory muscle Training Group
- Conventional Breathing Exercise Group (Active Comparator): Breathing Ex: Pursed lip Breathing, Diaphragmatic breathing ex, incentive spirometer
  Interventions: Other: Conventional Breathing Exercise Group

INTERVENTIONS:
Other: Resistive Expiratory muscle Training Group — Mild Resistive Expiratory Technique [Expiratory Muscle Strength Training (EMST150)- six-week training protocol approximately 20 min per day] The EMST requires the participant to forcibly blow into the device for 5 seconds with sufficient pressure to open the one-way valve. Each "blow" is one repetition. The device will be set at a resistance of 30 cmH2O. Participants will be instructed to complete five sets of five repetitions (total of 25 times and approximately 20 minutes per day), any five days per week, for six weeks. Whole exercise will be done in sitting position. Rest between repetitions will be given according to comfort level of patient.
  Arms: Resistive Expiratory muscle Training Group
Other: Conventional Breathing Exercise Group — Breathing Exercises: (approximately 20 minutes per day)
  ● Pursed lip breathing: (Sit with your back straight. Inhale through your nose for two seconds. Purse your lips like you're blowing on hot food and then breathe out slowly, taking twice as long to exhale as you took to breathe in. 4-5 times a day)
  ● Diaphragmatic breathing: (Lie on your back on a flat surface, knees bent and head supported. Use pillow under knees to support your legs. Breathe in slowly through your nose Tighten your stomach muscles, letting them fall inward as you exhale through pursed lips. Practice this exercise 5-10 minutes about 3-4 times per day).
  ● Incentive spirometer: (Hold in an upright position. Breathe in slowly and as deeply as possible. Hold your breath as long as possible (at least for 5 seconds). Then exhale slowly Rest for a few seconds and at least 10 times every hour)
  Arms: Conventional Breathing Exercise Group

SUMMARY:
* To determine effects of resistive expiratory muscle training on pulmonary functions in Chronic obstructive pulmonary disease (COPD) patients
* To determine effects of resistive expiratory muscle training on maximum expiratory pressure in COPD patients
* To determine effects of resistive expiratory muscle training on quality of life in COPD patients

ELIGIBILITY:
Inclusion Criteria:

* COPD patients (GOLD criteria - moderate, moderately severe)
* Borg scale < 4

Exclusion Criteria:

* Patients with Orthopedic disease
* Neurological disease,
* Cognitive impairment (Mini-Mental State Examination < 22) ,
* Heart diseases,
* Pulmonary fibrosis
* Obstructive sleep apnea syndrome.
* Acute and chronic infections

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Maximum expiratory pressure | 6 weeks
  Maximum expiratory pressure (MEP) measures the maximum positive pressure that can be generated from one expiratory effort starting from total lung capacity (TLC) . Changes will be assessed from the baseline and at the end of the intervention after 6 weeks
St George's Respiratory Questionnaire | 6 Week
  This is a specific respiratory instrument developed for patients with COPD. Its validity, reproducibility and response to change over time have been demonstrated. It has three components: symptoms, activity and impact. The responses to the items can be aggregated into an overall score and three sub-scores for symptoms, activity and impact in the range 0-100%. Higher scores indicate a poorer quality of life).Changes will be assessed from the baseline and at the end of the intervention after 6 weeks
Forced Expiratory Volume in 1 second (FEV1) | 6 Week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 6 week
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters.
Peak Expiratory Flow (PEF) | 6 Week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.
Volume of Lungs inflation | 6 week
  The incentive spirometer is a device that encourages patients with visual and other positive feedback, to maximally inflate their lungs and sustain that inflation. It is a common mode of postoperative respiratory therapy and involves deep breathing facilitated by a simple mechanical device. Maximal volume of lung inflation is thought to open collapsed alveoli and thereby prevent and resolve atelectasis. When all three balls reached their column tops, it indicated that the subject was able to generate inspiratory airflow of 1200 ml/ml. When only two balls reached their column tops, it indicated that the subject generated 900 ml/min. When only one ball reached their column tops, it indicated that the subject could only generate 600 ml/min. Changes will be assessed from the baseline and at the end of the intervention after 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Holy Family Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No